CLINICAL TRIAL: NCT03077347
Title: The Effects of Transcranial Direct Current Stimulation on the Neuronal Mechanisms of Cognitive Control in Schizophrenia
Brief Title: The Effects of tDCS on the Neuronal Mechanisms of Cognitive Control in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Per request of the study PI (fyi: NOT due to adverse events).
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1016455
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Transcranial Direct Current Stimulation; tDCS; Cognitive Control; fMRI; Dorsolateral Prefrontal Cortex
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Sham Stimulation followed by Direct Current Stimulation or Vice-Versa
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sham Followed by Experimental Stimulation (Other): Sham stimulation administered followed by 24-48 hour washout, then experimental stimulation.
  Experimental Intervention. 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex Placebo Comparator. 1 minute of 2 mA direct current stimulation over the dorsolateral prefrontal cortex followed by 19 minutes of sham stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation
- Experimental Stimulation Followed by Sham (Other): Experimental stimulation administered followed by 24-48 hour washout, then sham stimulation.
  Experimental Intervention. 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex Placebo Comparator. 1 minute of 2 mA direct current stimulation over the dorsolateral prefrontal cortex followed by 19 minutes of sham stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, saline-soaked electrodes are temporary affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (~20 minutes) to stimulate the targeted brain area (e.g. the DLPFC). To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation.
  Other Names: tDCS

SUMMARY:
The purpose of this study is to better understand the neural correlates of cognitive control (CC) deficits in schizophrenia and determine how these mechanisms can be modulated by transcranial direct current stimulation (tDCS). CC is a critical neurocognitive process that is required for flexible, directed thought and action based on goals and intentions. Identifying and developing paradigms to improve CC is therefore a mental health priority. Current theories of CC postulate that recruitment of the dorsolateral prefrontal cortex (DLPFC) is essential for this process by maintaining high-level information that it can then use to orchestrate patterns of activation in other brain networks to support optimal performance. tDCS is a safe, noninvasive method of modulating regional brain excitability via brief (15-20 m) application of a weak (1-2 mA) current. The goal of the proposed experiments is to combine tDCS with functional magnetic resonance imaging (fMRI) to test the hypotheses that 1) acute tDCS over the DLPFC can improve performance during a CC task (the dot pattern expectancy (DPX) variant of the AX-Continuous Performance Task) in schizophrenia patients and healthy control subjects, and 2) acute tDCS over the DLPFC can increase recruitment of the DLPFC during the DPX. Effects of tDCS on brain functional connectivity (during CC as well as during the resting state) will also be examined, as well as effects on an episodic memory task. The current study will be the first to use functional magnetic resonance imaging (fMRI) to examine the effects of tDCS on the neuronal mechanisms of CC in schizophrenia, and has potentially important implications for therapeutic development for this treatment refractory yet disabling aspect of the illness.

ELIGIBILITY:
Inclusion Criteria

* Sufficient English literacy so as to be able to understand and complete cognitive tasks.
* The ability to give valid informed consent.
* Diagnosis of schizophrenia, schizophreniform or schizoaffective disorder (for patient group)
* Stable outpatient or partial hospital status (for patient group)

Exclusion Criteria

* Psychiatric medication changes in the prior month (for patient group)
* No psychiatric medication changes anticipated in the upcoming month (for patient group)
* Intelligence Quotient (IQ) < 70; IQ will be measured by administering the Wechsler Abbreviated Scale of Intelligence (WASI) test.
* People under the age of 18
* Pregnant Women
* Prisoners
* Pacemakers
* Implanted brain stimulators
* Implanted defibrillator
* Metallic implants
* Skin damage or skin conditions such as eczema at the sites where electrodes will be placed
* Dreadlocks or other hair styles hindering the placement of tDCS electrodes
* Cranial pathologies
* Head trauma
* Epilepsy
* Mental retardation
* Neurological disorders
* Uncorrected vision problems that would hinder cognitive testing (this also pertains to subjects with color blindness in tasks where discriminating colored objects/items is necessary for successful performance).
* Other than nicotine, no subjects reporting substance dependence in the past six months and no substance abuse in the past month

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Carter, M.D., Study Director — University of California, Davis
Locations (1):
- Imaging Research Center, University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Select data from this study may be submitted to the National Institute of Mental Health Data Archive (NDA). NDA is a data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying mental illness to collect and share de-identified information with each other. The data repository is accessible only to qualified investigators. All subject data will be de-identified (subject names will not be used) and each subject will have a separate identifier called a Global Unique Identifier (GUID) to remove any possibility that "the identities of the subjects cannot be readily ascertained or otherwise associated with the data by the repository staff or secondary data users" (45 Code of Federal Regulations, 46.102).

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham First, Then Experimental Stimulation: Sham: Very brief 2 mA constant stimulation (~1 minute). Experimental: 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex.
  Transcranial Direct Current Stimulation: In tDCS, saline-soaked electrodes are temporary affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (~20 minutes) to stimulate the targeted brain area (e.g. the DLPFC). To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation.
  In this arm, sham was given first, followed by a washout period of 24-48 hours, followed by the experimental TDCS stimulation.
- Experimental Stimulation First, Then Sham: Experimental: 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex Sham: Very brief 2 mA constant stimulation (~1 minute).
  Transcranial Direct Current Stimulation: In tDCS, saline-soaked electrodes are temporary affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (~20 minutes) to stimulate the targeted brain area (e.g. the DLPFC). To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation.
  In this arm, the experimental TDCS stimulation was given first, followed by a washout period of 24-48 hours, followed by sham.
Period: Sham Stimulation (1-20 Minutes)
Arm/Group | Sham First, Then Experimental Stimulation | Experimental Stimulation First, Then Sham
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Washout (24-48 Hours)
Arm/Group | Sham First, Then Experimental Stimulation | Experimental Stimulation First, Then Sham
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Experimental Stimulation (1-20 Minutes)
Arm/Group | Sham First, Then Experimental Stimulation | Experimental Stimulation First, Then Sham
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Followed by Experimental Stimulation: This study will use a crossover design. In this arm, the sham stimulation is followed by a 24-48 hour washout period, followed by experimental stimulation.
  Experimental Intervention: 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex Sham: 1 minute fo 2 mA direct current stimulation over the dorsolateral prefrontal cortex
  Transcranial Direct Current Stimulation: In tDCS, saline-soaked electrodes are temporary affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (~20 minutes) to stimulate the targeted brain area (e.g. the DLPFC). To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation. The study will use a crossover design.
  To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation.
  I
- Experimental Stimulation Followed by Sham: This study will use a crossover design. In this arm, the experimental stimulation is followed by a 24-48 hour washout period, followed by sham stimulation.
  Experimental Intervention: 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex Sham: 1 minute fo 2 mA direct current stimulation over the dorsolateral prefrontal cortex
  Transcranial Direct Current Stimulation: In tDCS, saline-soaked electrodes are temporary affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (~20 minutes) to stimulate the targeted brain area (e.g. the DLPFC). To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation. The study will use a crossover design.
  To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation.
- Total: Total of all reporting groups
Arm/Group | Sham Followed by Experimental Stimulation | Experimental Stimulation Followed by Sham | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (3) | 21 (3) | 21 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Dorsolateral Prefrontal Cortex Response
Description: Blood oxygen level-dependent response of the dorsolateral prefrontal cortex during a cognitive control task (Dot-Probe Expectancy Task)
Time Frame: Assessment will begin immediately following stimulation and last for up to an hour.
Measure: Mean (Standard Deviation); unit: beta weights of DLPFC fMRI activations
Groups:
- Sham Stimulation: To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute). Subjects usually cannot discern the difference between the sham and experimental stimulation protocols due to habituation.
- Experimental Stimulation: 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex
Arm/Group | Sham Stimulation | Experimental Stimulation
Number analyzed (Participants) | 6 | 6
beta weights of DLPFC fMRI activations | 1.46 (.76) | 1.49 (2.08)

2. Primary Outcome: Behavioral Response
Description: Cognitive control-related performance (d-prime context) associated with the task (Dot-Probe Expectancy Task).
  The d-prime context index was calculated by computing a d-prime index from hits on AX trials and false alarms on BX trials as Z(H) - Z(F), with H representing hits on AX trials, F representing false alarms on BX trials, and Z representing the z-transform of a value.
  Positive d-prime values indicate more cognitive control, and negative values indicate less cognitive control.
Time Frame: Assessment will begin immediately following stimulation and last for up to an hour.
Measure: Mean (Standard Deviation); unit: d-prime context
Groups:
- Sham Stimulation: Sham: To control for placebo effects, the study will utilize a sham stimulation protocol that consists of very brief constant stimulation (~1 minute 2 mA).
- Experimental Stimulation: Experimental. 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex
Arm/Group | Sham Stimulation | Experimental Stimulation
Number analyzed (Participants) | 6 | 6
d-prime context | 3.35 (.25) | 3.12 (.91)

ADVERSE EVENTS:
Time Frame: 3 days
Groups:
- Sham Stimulation: The sham stimulation protocol consists of very brief constant stimulation (~1 minute 20 mA).
- Experimental Stimulation: 20 minutes 2 mA transcranial direct current stimulation.
Arm/Group | Sham Stimulation | Experimental Stimulation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03077347/Prot_001.pdf